CLINICAL TRIAL: NCT02107976
Title: Famine From Feast: Linking Vitamin C, Red Blood Cell Fragility, and Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 140060; 14-DK-0060
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-08-20

CONDITIONS: Diabetes Type 2
Keywords: Diabetes; Red Blood Cells; Vitamin C; Plasma Vitamin C Levels
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vitamin E; Ascorbic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage 1 (Experimental): Inpatient admission to NIH CC, consisting of euglycemic period with serial blood and urine sampling followed by hyperglycemic period (induced with high-carbohydrate diet; diabetic subjects only) with serial blood and urine sampling.
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Vitamin C
- Stage 2 (Experimental): Inpatient admission to NIH CC after at least 8 weeks of vitamin C and vitamin E supplementation. Testing periods include: euglycemic period with serial blood and urine sampling followed by hyperglycemic period (induced with high-carbohydrate diet; diabetic subjects only) with serial blood and urine sampling.
  Interventions: Dietary Supplement: Vitamin E; Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin E — 400 IU per day after discharge, for a minimum of 8 weeks between Stage 1 and Stage 2
Dietary Supplement: Vitamin C — 500mg twice a day after discharge, for a minimum of 8 weeks between Stage 1 and Stage 2

SUMMARY:
Diabetes type two is a debilitating disease that leads to chronic morbidity such as accelerated microvascular disease. Accelerated microvascular disease may produce blindness, end stage renal disease, myocardial infarction, stroke, and limb ischemia. Strategies to prevent or delay microvascular disease have the potential to improve the lives of millions and prevent catastrophic illness. The major focus of prevention of microvascular disease in diabetes has been on the endothelium and its role in protection of blood vessels. An unexpected means to prevent microvascular disease in diabetes may be coupled to the function of vitamin C in red blood cells (RBCs) of diabetic subjects. Based on new and emerging data, vitamin C concentrations in RBCs may be inversely related to glucose concentrations found in diabetes. Based on animal data, we hypothesize that RBCs with low vitamin C levels may have decreased deformability, leading to slower flow in capillaries and microvascular hypoxia, the hallmark of diabetic microangiopathy. Low vitamin C concentrations in RBCs of diabetic subjects may be able to be increased, by using vitamin C supplements. Findings in animals may not accurately reflect effects in humans because of species differences in mechanisms of vitamin C entry into RBCs. Therefore, clinical research is essential to characterize vitamin C physiology in RBCs of diabetic subjects. In this protocol we will investigate physiology of vitamin C in RBCs of diabetic subjects as a function of glycemia, without vitamin C supplementation (stage 1) and with vitamin C supplementation (stage 2). We will screen type II diabetic subjects on insulin and/or oral hypoglycemic medication(s) and select those with hemoglobin A1C concentrations of less than or equal to 12%. Selected subjects may be hospitalized twice, each time for approximately one week. The primary objective of the first hospitalization (stage 1) will be to evaluate the effect of hyperglycemia on vitamin C RBC physiology regardless of baseline vitamin C concentrations (without any vitamin C supplementation). The second hospitalization (stage 2) investigates the effect (if any) of vitamin C supplementation to changes in RBC physiology during euglycemic and hyperglycemic states. As inpatients, subjects will have two venous sampling periods each of approximately 24 hours. On admission, subjects may be fitted with continuous glucose monitors (CGMs), oral hypoglycemic agents will be discontinued, and basal-bolus insulin regimen initiated. Insulin doses will be clinically determined and titrated to achieve euglycemia (fasting and pre-meal glucoses <140mg/dl) prior to the first sampling period (euglycemic sampling). The first sampling period will be performed under conditions of euglycemic control for 24 hours. The second sampling period will be performed under controlled hyperglycemia induced by withholding basal and bolus insulin and providing a high carbohydrate load diet (70-75% carbohydrate). Correction-scale insulin will be provided for glucoses >350-400mg/dl. Hyperglycemia will not exceed 9 hours, and will be reversed by reinstituting insulin.

During the two sampling periods, samples will be withdrawn via venous catheter for RBC deformability, vitamin C concentrations and other related research studies. Following completion of stage 1, subjects considered for participation in stage 2 will be provided a prescription for vitamin C 500mg twice daily. Given that vitamin C and vitamin E are related antioxidants, and that both vitamins appear to be associated with RBC rigidity, diabetic subjects may also be given a prescription for 400 international units (IU) of vitamin E (RRR alpha tocopherol) daily. Subjects will continue vitamin C and E supplementation for a minimum of 8 weeks depending on RBC vitamin C concentrations. To evaluate any effect of vitamin E supplementation, plasma and RBC vitamin E levels may be measured concurrently with vitamin C levels during various phases of stages 1 and 2. All subjects will be seen as outpatients at biweekly or monthly intervals with regular measurement of plasma and RBC vitamin C concentrations. Target RBC vitamin C concentration >30uM is required prior to stage 2 inpatient sampling studies. Vitamins C and E supplementation will be discontinued upon inpatient admission for stage 2. Risk of both vitamin supplements are minimal as both supplementation doses are safe. Outcomes are to measure RBC rigidity and vitamin concentrations before and after supplementation. After a minimum of 8 weeks (depending on RBC vitamin C levels), subjects will be hospitalized again, and sampling repeated as described. In this manner, each subject serves as his/her own control, and deformability of red blood cells can be determined in relation to glycemia and to vitamin C concentrations in RBCs and plasma.

DETAILED DESCRIPTION:
Diabetes type two is a debilitating disease that leads to chronic morbidity such as accelerated microvascular disease. Accelerated microvascular disease may produce blindness, end stage renal disease, myocardial infarction, stroke, and limb ischemia. Strategies to prevent or delay microvascular disease have the potential to improve the lives of millions and prevent catastrophic illness. The major focus of prevention of microvascular disease in diabetes has been on the endothelium and its role in protection of blood vessels. An unexpected means to prevent microvascular disease in diabetes may be coupled to the function of vitamin C in red blood cells (RBCs) of diabetic subjects. Based on new and emerging data, vitamin C concentrations in RBCs may be inversely related to glucose concentrations found in diabetes. Based on animal data, we hypothesize that RBCs with low vitamin C levels may have decreased deformability, leading to slower flow in capillaries and microvascular hypoxia, the hallmark of diabetic microangiopathy. Low vitamin C concentrations in RBCs of diabetic subjects may be able to be increased, by using vitamin C supplements. Findings in animals may not accurately reflect effects in humans because of species differences in mechanisms of vitamin C entry into RBCs. Therefore, clinical research is essential to characterize vitamin C physiology in RBCs of diabetic subjects. In this protocol we will investigate physiology of vitamin C in RBCs of diabetic subjects as a function of glycemia, without vitamin C supplementation (stage 1) and with vitamin C supplementation (stage 2). We will screen type II diabetic subjects on insulin and/or oral hypoglycemic medication(s) and select those with hemoglobin A1C concentrations of <= 12%. To investigate how response to the nutritional interventions in individuals with diabetes varies from normal, nondiabetic controls will also be recruited and studied. Selected subjects will be hospitalized twice, each time for approximately one week. The primary objective of the first hospitalization (stage 1) will be to evaluate the effect of hyperglycemia on vitamin C RBC physiology regardless of baseline vitamin C concentrations (without any vitamin C supplementation). The second hospitalization (stage 2) investigates the effect (if any) of vitamin C supplementation to changes in RBC physiology during periods of normal (euglycemic) and elevated (hyperglycemic) glucose concentrations. As inpatients, subjects will have two venous sampling periods each of approximately 24 hours.

On admission, subjects may be fitted with continuous glucose monitors (CGMs), subjects will be transitioned to an individualized inpatient diabetes regimen determined by investigators, based on pre-admission diabetes regimen and glycemic control. For participants with diabetes, the inpatient diabetes regimen will be titrated to achieve euglycemia (fasting and pre-meal glucoses <140mg/dl) prior to the first sampling period (euglycemic sampling). The first sampling period will be performed under conditions of euglycemic control for 24 hours. The second sampling period will be performed under controlled hyperglycemia induced by decreasing doses of the diabetes regimen and providing a high carbohydrate load diet (70-75% carbohydrate). Correction-scale insulin will be provided for glucoses >350-400mg/dl. Hyperglycemia will not exceed 9 hours and will be reversed by reinstituting insulin. For nondiabetic controls, an oral glucose tolerance test (75 grams dextrose) will be administered on admission. Controls will receive the same metabolic diets and undergo the sampling schedule as the cohort with diabetes. During the two sampling periods, samples will be withdrawn via venous catheter for RBC deformability, vitamin C concentrations and other related research studies. Following completion of stage 1, subjects considered for participation in stage 2 will be provided a prescription for vitamin C 500mg twice daily. Given that vitamin C and vitamin E are related antioxidants, and that both vitamins appear to be associated with RBC rigidity, diabetic subjects may also be given a prescription for 400 international units (IU) of vitamin E (RRR alpha tocopherol) daily. Subjects will continue vitamin C and E supplementation for a minimum of 8 weeks depending on RBC vitamin C concentrations. To evaluate any effect of vitamin E supplementation, plasma and RBC vitamin E levels may be measured concurrently with vitamin C levels during various phases of stages 1 and 2. All subjects will be seen as outpatients at biweekly or monthly intervals with regular measurement of plasma and/or RBC vitamin C concentrations. Target RBC vitamin C concentration >30uM is required prior to stage 2 inpatient sampling studies. Vitamins C and E supplementation will be discontinued upon inpatient admission for stage 2. Risk of both vitamin supplements are minimal as both supplementation doses are safe. Outcomes are to measure RBC rigidity and vitamin concentrations before and after supplementation. After a minimum of 8 weeks (depending on RBC vitamin C levels), subjects will be hospitalized again, and sampling repeated as described. In this manner, each subject serves as his/her own control, and deformability of red blood cells can be determined in relation to glycemia and to vitamin C concentrations in RBCs and plasma. Subjects will be required to consume standardized meals during inpatient stays. All meals will be prepared by the NIH Clinical Center Metabolic Kitchen. To avoid obscuring plasma vitamin C changes that may result from hyperglycemia, dietary vitamin C content will be approximately 30-35 mg per meal. Additionally, to avoid confounding vitamin E measurements, diets will provide approximately 6 mg alpha tocopherol per day. Standardized meals at the 2nd inpatient admission will be provided to match what was consumed by the subject at their 1st inpatient admission.

ELIGIBILITY:
* INCLUSION CRITERIA:

Stage 1

* Male or female 18-65 years old, able to give informed consent.
* Diabetes type 2 HgA1C <= 12% on insulin and/or oral hypoglycemic agents or nondiabetic without any prior history or diagnosis of diabetes.
* In general good health with no other significant illness.
* Mild concomitant disease such as mild hypothyroidism (TSH <10) is acceptable.
* Blood pressure with or without medication <160/90 mmHg with no known significant target organ damage (end organ damage includes the following: proliferative retinopathy, serum creatinine >1.5 or EGFR < 55 mL/min, symptomatic ischemic heart disease, severe congestive heart failure, advanced peripheral vascular disease.
* Willingness to use effective contraceptive methods such as barrier method for the duration of study (female subjects).

Stage 2

Above criteria with addition of RBC vitamin C concentration >30 uM prior to inpatient studies.

EXCLUSION CRITERIA:

Stage 1 and 2

* Diabetic type 1 subjects will be excluded due to the possibility of ketosis and hemodynamic instability with lack of insulin.
* Any subjective or objective evidence of microangiopathy such as history of claudication, symptomatic peripheral vascular disease, symptomatic coronary artery disease, stroke, retinopathy, nephropathy (serum creatinine >1.5 or EGFR < 55 mL/min).
* Diabetic subjects with retinopathy to avoid accelerated retinopathy with hyperglycemia.
* Concomitant disease such as severe heart failure, severe liver disease (transaminases > 3 times normal), or severe systemic disease of any sort.
* Pregnancy, breastfeeding.
* History of diabetic ketoacidosis or hyperosmolar coma.
* Subjects with clear evidence of non-compliance with protocol/study instructions.
* Subjects who are unwilling or lack capacity to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Change in RBC deformability half maximal shear stress (SS0.5) from stage 1 to stage 2 | End of stage 2
  RBC SS0.5 is another measure of RBC deformability hypothesized to increase after dietary vitamin C and vitamin E supplmentation in diabetic subjects.
Change in RBC deformability maximum elongation indices (EImax) from stage 1 to stage2 | End of stage 2
  RBC EImax is hypothesized to increase in people with diabetes following vitamin C and vitamin E dietary supplementation.
Change in RBC deformability elongation indices (EI) from stage 1 to stage 2 | End of stage 2
  Red blood cell (RBC) deformability measures the ability of the RBC to change shape upon entering into capillaries. RBC deformability is vital to RBC function and impaired deformability adversely affects capillary perfusion. Vitamins C and E supplementation is hypothesized to increase RBC deformability EI in people with diabetes.

SECONDARY OUTCOMES:
Change in RBC deformability maximum elongation indices (EImax) | before and afterhyperglycemic intervention during stage 1
  Examine the effect of hyperglycemia on RBC EImax
Change in RBC deformability elongation indices | before and after hyperglycemicintervention during stage 1
  Examines the effect of hyperglycemia on RBC EI
Change in RBC deformability half-maximal shear stress (SS0.5) | before and afterhyperglycemic intervention during stage 1
  Examine the effect of hyperglycemia on RBC SS0.5
Change in vitamin C concentration in plasma | from stage 1 to stage 2
  Determine whether at least 8 weeks of dietary supplementation with vitamin C increases plasma vitamin C levels
Change in vitamin C concentration in urine | from stage 1 to stage 2
  Determine whether at least 8 weeks of dietary supplementation with vitamin C increases urine vitamin C levels
Change in vitamin C concentration in RBC | from stage 1 to stage 2
  Determine whether at least 8 weeks of dietary supplementation with vitamin C increases RBC vitamin C levels
Change in vitamin C concentrations in plasma | before and after hyperglycemic interventionduring stage 1
  Examine the effect of a transient hyperglycemic period on plasma vitamin C concentrations
Change in vitamin C concentrations in RBC | before and after hyperglycemic interventionduring stage 1
  Examine the effect of a transient hyperglycemic period on RBC vitamin C concentrations
Change in vitamin C concentrations in urine | before and after hyperglycemic interventionduring stage 1
  Examine the effect of a transient hyperglycemic period on urine vitamin C concentrations
Change in vitamin E concentration in plasma | from stage 1 to stage 2
  Examine the effect of at least 8 weeks of dietary vitamin E supplementation on plasma vitamin E concentrations
Change in vitamin E concentration in RBC | from stage 1 to stage 2
  Examine the effect of at least 8 weeks of dietary vitamin E supplementation on RBC vitamin E concentrations
Change in plasma isoprostane concentrations | from stage 1 to stage 2
  Examine the effect of at least 8 weeks of dietary vitamin C and E supplementation on plasma isoprostane concentrations
Change in plasma isoprostane concentrations | before and after hyperglycemic interventionduring stage 1
  Examine the effect of a transient hyperglycemic period on plasma isoprostane concentrations
Change in urine isoprostane concentrations | from stage 1 to stage 2
  Examine the effect of at least 8 weeks of dietary vitamin C and E supplementation on urine isoprostane concentrations
Change in urine isoprostane concentrations | before and after hyperglycemic interventionduring stage 1
  Examine the effect of a transient hyperglycemic period on urine isoprostane concentrations
Change in SF-36 health related quality of life survey | from stage 1 to stage 2
  Examine whether self-reported quality of life improves with at least 8 weeks of vitamin C and E dietary supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Ifechukwude C Ebenuwa, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ali SM, Chakraborty SK. Role of plasma ascorbate in diabetic microangiopathy. Bangladesh Med Res Counc Bull. 1989 Dec;15(2):47-59. PMID 2629696
- [Background] Baskurt OK, Hardeman MR, Uyuklu M, Ulker P, Cengiz M, Nemeth N, Shin S, Alexy T, Meiselman HJ. Comparison of three commercially available ektacytometers with different shearing geometries. Biorheology. 2009;46(3):251-64. doi: 10.3233/BIR-2009-0536. PMID 19581731
- [Background] Beckman JA, Creager MA, Libby P. Diabetes and atherosclerosis: epidemiology, pathophysiology, and management. JAMA. 2002 May 15;287(19):2570-81. doi: 10.1001/jama.287.19.2570. PMID 12020339
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-DK-0060.html